CLINICAL TRIAL: NCT06027281
Title: Psychiatric, Social and Sexual Consequences of Female Genital Mutilation on Married Women
Brief Title: Consequences of Female Genital Mutilation on Married Women.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Gamil Kamel, Principal investigator, Assiut University
Other Study IDs: Consequences of FGM
Record Dates: First submitted 2023-02-18; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Female Genital Mutilation
Keywords: Psychiatric; Social; Sexual; Married
MeSH Terms: conditions — Coitus | interventions — Psychiatric Status Rating Scales; MMPI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Married women who had female genital mutilation
  Interventions: Other: Hamilton depression rating scale (HDRS); Other: Hamilton anxiety rating scale (HARS); Other: Mini international neuropsychiatric interview (MINI); Other: Minnesota Multiphasic personality Inventory (MMPI); Other: The Symptom Check-List-90-R (SCL-90-R); Other: Socioeconomic scale (A.El Gilany, A.El Wehady and M.El Wasify); Other: The female sexual function index (FSFI)
- Married women who didn't have female genital mutilation
  Interventions: Other: Hamilton depression rating scale (HDRS); Other: Hamilton anxiety rating scale (HARS); Other: Mini international neuropsychiatric interview (MINI); Other: Minnesota Multiphasic personality Inventory (MMPI); Other: The Symptom Check-List-90-R (SCL-90-R); Other: Socioeconomic scale (A.El Gilany, A.El Wehady and M.El Wasify); Other: The female sexual function index (FSFI)

INTERVENTIONS:
Other: Hamilton depression rating scale (HDRS) — Hamilton depression scale (HDRS) is the most commonly used instrument for assessing symptoms of depression.
Other: Hamilton anxiety rating scale (HARS) — Hamilton anxiety rating scale (HARS) is a 14-item clinician-rated measure of the severity of perceived anxiety symptoms.
Other: Mini international neuropsychiatric interview (MINI) — The Mini International Neuropsychiatric Interview (MINI) was designed as a brief structured diagnostic interview for the major psychiatric disorders in DSM-III-R, DSM-IV and DSM-5 and ICD-10.
Other: Minnesota Multiphasic personality Inventory (MMPI) — The Minnesota Multiphasic Personality Inventory (MMPI) is used to assess personality traits and psychopathology.
Other: The Symptom Check-List-90-R (SCL-90-R) — The Symptom Check-List-90-R (SCL-90-R) is a widely used psychological status symptom inventory.
Other: Socioeconomic scale (A.El Gilany, A.El Wehady and M.El Wasify) — An Arabic version of the socioeconomic scale consisted of four dimensions, namely, level of education, employment, total family monthly income, and lifestyle of the family.
Other: The female sexual function index (FSFI) — The female sexual function index is a brief multidimensional scale for assessing sexual function in women.

SUMMARY:
To assess psychiatric, social and sexual consequences of female genital mutilation on married women.

DETAILED DESCRIPTION:
World Health Organization (WHO) defined female genital mutilation (FGM) as ''all procedures that involve partial or total removal of the external female genitalia, or other injury to the female genital organs for non-medical reasons.

Many countries throughout the globe perform it: Western, Eastern, and North-Eastern Africa, particularly Egypt and Ethiopia, and in parts of Asia and the Middle East (nearly half of its cases are in Egypt and Ethiopia).

Moreover, the prevalence of girls and women with FGM/C is also rising in Western countries due to migration flows.

The adverse physical consequences of female genital mutilation/cutting (FGM/C) have been thoroughly investigated and documented. Yet, we know little about the adverse mental health consequences of the practice.

Also, few systematic reviews have addressed the impact of the practice on psycho-social well-being, and there is limited understanding of what these consequences might consist.

Throughout Egypt, many studies have been conducted to determine the pattern and prevalence of FGM, but those studied the risks of FGM and its effect on women's sexual life are scare.

ELIGIBILITY:
Inclusion Criteria:

* Married females aged 18-50 years.

Exclusion Criteria:

* Women who have any chronic disease as diabetes or hypertension.
* Women who have any physical or mental handicap.
* Women who have any psychiatric disorder prior to marriage.
* Women who refuse participation in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Married women aged 18-50 years old.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton depression rating scale (HDRS) | From 10 to 15 minutes
  To determine severity of anxiety.
Hamilton anxiety rating scale (HARS) | From 10 to 15 minutes
  To determine severity of anxiety.
Screening for psychiatric symptoms. | From 20 to 30 minutes
  Mini international neuropsychiatric interview (MINI)
Screening for psychiatric symptoms. | From 45 to 60 minutes
  Minnesota Multiphasic personality Inventory (MMPI)
Determination of socioeconomic class of the family. | From 15 to 20 minutes
  Family socioeconomic status scale (revised version 2019)
Screening for female sexual dysfunction. | From 15 to 20 minutes
  The female sexual function index (FSFI)

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Gamil Kamel, Study Director — Assiut University; Wageh Abd El Nasser Hassan, PhD, Principal Investigator — Assiut University; Mostafa Mahmoud Elnoamany, PhD, Principal Investigator — Assiut Univesity

REFERENCES:
- [Result] Abdalla SM, Galea S. Is female genital mutilation/cutting associated with adverse mental health consequences? A systematic review of the evidence. BMJ Glob Health. 2019 Jul 15;4(4):e001553. doi: 10.1136/bmjgh-2019-001553. eCollection 2019. PMID 31406589
- [Result] O'Neill S, Pallitto C. The Consequences of Female Genital Mutilation on Psycho-Social Well-Being: A Systematic Review of Qualitative Research. Qual Health Res. 2021 Jul;31(9):1738-1750. doi: 10.1177/10497323211001862. Epub 2021 Jun 8. PMID 34098783
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Thompson E. Hamilton Rating Scale for Anxiety (HAM-A). Occup Med (Lond). 2015 Oct;65(7):601. doi: 10.1093/occmed/kqv054. No abstract available. PMID 26370845
- [Result] Williams JB. Standardizing the Hamilton Depression Rating Scale: past, present, and future. Eur Arch Psychiatry Clin Neurosci. 2001;251 Suppl 2:II6-12. doi: 10.1007/BF03035120. PMID 11824839
- [Result] Pettersson A, Modin S, Wahlstrom R, Af Winklerfelt Hammarberg S, Krakau I. The Mini-International Neuropsychiatric Interview is useful and well accepted as part of the clinical assessment for depression and anxiety in primary care: a mixed-methods study. BMC Fam Pract. 2018 Jan 24;19(1):19. doi: 10.1186/s12875-017-0674-5. PMID 29368585
- [Result] van Vliet IM, de Beurs E. [The MINI-International Neuropsychiatric Interview. A brief structured diagnostic psychiatric interview for DSM-IV en ICD-10 psychiatric disorders]. Tijdschr Psychiatr. 2007;49(6):393-7. Dutch. PMID 17614093
- [Result] Floyd AE, Gupta V. Minnesota Multiphasic Personality Inventory. 2023 Apr 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557525/ PMID 32491457
- [Result] Schmitz N, Hartkamp N, Kiuse J, Franke GH, Reister G, Tress W. The Symptom Check-List-90-R (SCL-90-R): a German validation study. Qual Life Res. 2000 Mar;9(2):185-93. doi: 10.1023/a:1008931926181. PMID 10983482